CLINICAL TRIAL: NCT03790007
Title: COMPARISON OF INTRAOPERATIVE TRANSVERSUS ABDOMINIS PLANE BLOCK, LOCAL ANESTHESIA APPLICATION TO THE PORT SITES AND INTRAPERITONEAL LOCAL ANESTHETIC APPLICATIONS IN POSTOPERATIVE PAIN MANAGEMENT IN LAPAROSCOPIC CHOLECYSTECTOMY PATIENTS
Brief Title: COMPARISON OF INTRAOPERATIVE LOCAL ANESTHETIC APPLICATIONS IN POSTOPERATIVE PAIN MANAGEMENT IN LAPAROSCOPIC CHOLECYSTECTOMY PATIENTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, asistant doctor, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ANIL ERGIN....
Record Dates: First submitted 2018-12-15; First posted 2018-12-31 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Pain
Keywords: laparoscopic cholecystectomy; postoperative pain relief; local anesthetic
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: 3 types of local anesthetic applying method will be compared
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Transversus Abdominis Plane Block (Active Comparator): Transversus abdominis plane block (10 cc / 10 cc, 0.5% bupivacaine to the right and left transversus abdominis muscle regions) will be applied.
  Interventions: Drug: Bupivacaine
- TROCHAR SITES LOCAL ANESTHETIC INJECTION (Active Comparator): local anesthetic injection (6 cc to subxiphoid and infraumbilical trocar sites, 4 cc instead of 2 cc, 0.5% bupivacaine solution to be applied)
  Interventions: Drug: Bupivacaine
- INTRAPERİTONEAL LOCAL ANESTHETIC SPREADING METHOD (Active Comparator): Intraperitoneal direct vision of the gallbladder excision area-periportal area under the direct injection of local anesthetic spraying process (percutaneous method injected into the periportal area 1: 1 diluted with 20 cc SF, 20 cc 0.5% bupivacaine solution total 40 cc spraying will be applied.
  Interventions: Drug: Bupivacaine
- CONTROL GROUP (No Intervention): group will be the control group and any of these methods will not be applied,

INTERVENTIONS:
Drug: Bupivacaine — In our study this local anesthetic agent will be applied for postoperative pain relief
  Other Names: marcaine
  Arms: INTRAPERİTONEAL LOCAL ANESTHETIC SPREADING METHOD; TROCHAR SITES LOCAL ANESTHETIC INJECTION; Transversus Abdominis Plane Block

SUMMARY:
Since 1987, laparoscopic cholecystectomy has become the standard procedure for gallbladder stones and lesions. Complications due to improvements in laparoscopy and increased surgical experience have decreased day by day, but there is still a problem in terms of postoperative pain management. Several pain management procedures have been tried to combat pain after laparoscopic cholecystectomy. The aim of this study is to decrease the length of hospital stay, to increase the comfort of the patient and to reduce the cost of treatment. Local anesthetic injection to port locations, intraperitoneal periportal local anesthetic injection ,Transversus Abdominis Plane Blok and without any local anesthetic application to the control group compared to the group's analgesic efficiency and to reduce the amount of analgesics needed, shorten the length of hospital stay and improve patient comfort.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy procedure will be performed in patients older than 18 years of age for the diagnosis of cholelithiasis. Laparoscopic cholecystectomy procedure will be performed.4 patients group will be formed Power: 0.80 and alpha: :0.05 The minimum number of samples determined for each group is n: 34 for each group. It will be determined. In our clinic, local anesthetic injections are performed routinely to the trocar areas in laparoscopic cholecystectomy operations. After endotracheal intubation at the beginning of the operation, after appropriate skin staining and sterile dressing, Transversus abdominis plane block (10 cc / 10 cc, 0.5% bupivacaine to the right and left transversus abdominis muscle regions) will be applied. to the second group local anesthetic injection (6 cc to subxiphoid and infraumbilical trocar sites, 4 cc instead of 2 cc, 0.5% bupivacaine solution) to be applied, in the third group intraperitoneal direct vision of the gallbladder area-periportal area under the direct injection of local anesthetic spraying process (percutaneous method injected into the periportal area 1: 1 diluted with 20 cc saline, 20 cc 0.5% bupivacaine solution total 40 cc spraying will be applied. The fourth group will be the control group and any of these methods will not be applied, the operation time and peroperative complications (pouch perforation etc.) will be recorded. Paracetamol 1 g + 1 mg / kg tramadol IV will be applied to all four groups as standard before extubation. Visual analogue scale (VAS) will be applied to all patients in the postoperative period. If VAS> 3 is still present, a dose of 1 mg / kg tramadol will be administered. Tenoxicam 1x1 IV will be applied to the patients on the 12th hour. All patients were postoperative; 1,2,4,6,12,24. VAS scores , patient satisfaction (0: never satisfied, 5: very satisfied) will be recorded. The group of patients will be determined according to the order of surgery. Pain scores of the patients will be performed by a physician who is not in the operation who does not know which group is taken. The patients included in the group will not be known to the patient by the pain scoring system and the study will be done as double blind. Patients will be randomized with this method.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who were admitted to the general surgery department with the diagnosis of cholelithiasis

Exclusion Criteria:

* Patients who need to undergo peroperative open cholecystectomy procedure.
* Patients with local anesthetic or NSAID allergy
* Patients in pregnancy
* Patients who are breastfeeding
* Patients with connective tissue disease
* Patients with malignancy in postoperative gallbladder pathological examination and patients with any malignancy diagnosis
* Patients with renal impairment, where the effect of using Marcain is unknown
* Cardiac disease
* Patients with hepatic impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Level of postoperative pain: visual analogue scale | 24 hours
  the level of the pain will be assessed using the VAS ( visual analogue scale) which is a psychometric response scale and the patient has to indicate a position along a continuous line between two end-points (no pain and maximum pain) that best reflects the intensity of their pain. The pain measurements will be done at 1,2,4,6,12,24 hours. Test is easy to obtain, reliable, valid and can detect changes of over time

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No